CLINICAL TRIAL: NCT06821256
Title: Efficacy and Safety of Transcranial dIrect Current stiMulation (tDCS) on Cerebellar Symptoms in Multiple System Atrophy-Cerebellar Variant (MSA-C) (STIM-MSA)
Brief Title: Efficacy and Safety of Transcranial dIrect Current stiMulation in Multiple System Atrophy-Cerebellar Variant
Acronym: STIM-MSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Roberto Erro, Principal Investigator, University of Salerno
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSA-STIM 01
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Multiple System Atrophy - Cerebellar Subtype (MSA-C)
Keywords: Multiple System Atrophy type C (MSA-C),; Transcranial direct current stimulation (tDCS)
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of the two arms and all will receive a sham-stimulation for 5 consecutive days/week (i.e.,Monday to Friday) and an active stimulation for 5 consecutive days/week (i.e., Monday to Friday). The order of the sham- vs active-stimulation will be also randomized within each arm. The active stimulation will consist of an anodal stimulation over the cerebellum area (2 cm under the inion, using a 7 × 5 cm sponge electrode), with the cathode being applied either to the right deltoid muscle (arm 1: cerebellar stimulation) or over the spinal lumbar enlargement (2 cm under T11; arm 2: cerebellar-spinal stimulation) using a sponge electrode of the same size as the anode. During anodal stimulation, a constant current of 2 mA will be applied for 20 minutes, as suggested by recently published consensus recommendations (Grimaldi et al, 2014). For the sham condition, the electrode placement will be the same as for the active stimulation, but the electric current
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomiziation, monitoring and data management will be performed locally. Randomization will be performed using an online list randomizer (random.org). The study coordinator will generate the random allocation sequence before enrollment. Then, one sub-investigator will perform clinical evaluations and another one will administer the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real tDCS group (Experimental): Partecipants receive anodal tDCS over the cerebellum area (2 cm under the inion, using a 7 × 5 cm sponge electrode), with the cathode being applied either to the right deltoid muscle (arm 1: cerebellar stimulation) or over the spinal lumbar enlargement (2 cm under T11; arm 2: cerebellar-spinal stimulation) using a sponge electrode of the same size as the anode for 5 days/week for 2 weeks
  Interventions: Device: Anodal transcranial direct current stimulation (a-tDCS)
- Sham group (Sham Comparator): Partecipants receive sham stimulation over the cerebellum area (2 cm under the inion, using a 7 × 5 cm sponge electrode), with the cathode being applied either to the right deltoid muscle (arm 1: cerebellar stimulation) or over the spinal lumbar enlargement (2 cm under T11; arm 2: cerebellar-spinal stimulation) using a sponge electrode of the same size as the anode for 5 days/week for 2 weeks
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation (a-tDCS) — tDCS is delivered by a battery-driven constant current stimulator throught a pair of saline soaked surface sponge electrodes. The active electrode (anode) is placed on the scalp over the over the cerebellum area (2 cm under the inion, using a 7 × 5 cm sponge electrode), with the cathode being applied either to the right deltoid muscle (arm 1: cerebellar stimulation) or over the spinal lumbar enlargement (2 cm under T11; arm 2: cerebellar-spinal stimulation) using a sponge electrode of the same size as the anode. Durng real stilumation a costant current of 2mA is applied for 20 minutes.
  Other Names: Active stimulation
  Arms: Real tDCS group
Device: Sham stimulation — For the sham condition the electrode placement is the same of active tDCS but the electric current is ramped down 5 seconds after the beginning of the stimulation
  Arms: Sham group

SUMMARY:
This is a double-blind, randomized, sham-controlled clinical trial that aim to verify the safety and the efficacy of anodal transcranial direct current stimulation (tDCS) cerebellar symptoms in Multiple System Atrophy type C (MSA).

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a progressive neurodegenerative disease for which, to date, no causal therapy is available, symptomatic treatment therefore playing a pivotal role in patient care (Fanciulli & Wenning, 2015). Unfortunately, there are very limited effective symptomatic treatments, especially for the cerebellar variant of MSA (MSA-C) which calls for the urgent need of developing alternative strategies to improve patients' disability and quality of life (QoL). An emergent approach to cerebellar disorders of various etiologies stands in the use of non-invasive brain stimulation (NIBS) techniques (Erro R et al., 2017), namely in the use of trans-cranial direct current stimulation (tDCS), to modulates neuronal excitability in a polarity-specific manner by delivering prolonged (up to 20-30 min) but weak (1-2 mA) currents to brain tissues via electrodes placed on the scalp (Stagg & Nitsche, 2011).

This project has been designed as a double-blinded, sham-controlled, cross-over trial with two independent arms to assess the feasibility and compare the efficacy of two different tDCS protocols. Sample size calculation has been calculated on preliminary unpublished results of our own research using tDCS in other atypical parkinsonisms (i.e., PSP) and we will accordingly recruit 15 patients for each arm of the study. Patients will be randomly assigned to one of the two arms and all will receive a sham-stimulation for 5 consecutive days/week (i.e.,Monday to Friday) and an active stimulation for 5 consecutive days/week (i.e., Monday to Friday). The order of the sham- vs active-stimulation will be also randomized within each arm. The active stimulation will consist of an anodal stimulation over the cerebellum area (2 cm under the inion, using a 7 × 5 cm sponge electrode), with the cathode being applied either to the right deltoid muscle (arm 1: cerebellar stimulation) or over the spinal lumbar enlargement (2 cm under T11; arm 2: cerebellar-spinal stimulation) using a sponge electrode of the same size as the anode. During anodal stimulation, a constant current of 2 mA will be applied for 20 minutes, as suggested by recently published consensus recommendations (Grimaldi et al, 2014). For the sham condition, the electrode placement will be the same as for the active stimulation, but the electric current will be ramped down 5 seconds after the beginning of the stimulation to make this condition indistinguishable from the experimental stimulation.

Before (T0), soon after the first week of the protocol (T1) and soon after the second week of the protocol (T2) all patients will be evaluated using 1) validated clinical scales for cerebellar disorders (SARA, ICARS) and 2) through the 8-m walking test (8MW); defined as the time needed to walk 8 m as quickly as possible but safely with any device but without the help of another person or wall. During the 8MW wearable sensors (OPAL) will be further used to collect objective measures of gait and balance. Finally, PROs will be collected by means of 1) the clinical global improvement measure (CGI-I) ranging from 1 (very much improved) to 7 (very much worse), with patients being asked to report their perceived improvement at T1 and T2; and 2) by two instruments for depicting change in QoL, namely the EuroQoL-5Dimensions, 3Levels (EQ-5D-3L) and the MSA-QoL (Schrag, Mov Disord 2007), both of which will be performed at T0, T1 and T2. Patients will be further asked whether they thought they were receiving real or sham stimulation at the end of the 2-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple system atrophy cerebellar variant according with the Movemente Disorder Society criteria (Wenning et al 2022)
* Ability to walk either indipendently or with a minimum support

Exclusion Criteria:

* Presence of electrical stimulators (for example, pacemaker, Deep Brain Stimulation, DBS)
* Difficult in understanding Italian language
* Presence of severe sensory deficits (for example, visual or hearing impairments)
* History of drug abuse
* History of severe psychiatric disorders
* History of transient ischemic attacks
* Cortical or sub-cortical vascular lesions
* Seizures or severe heart problems and previous neurosurgical operations
* Pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 1 week and two weeks follow in motor symptoms as assessed with sensor recordings (OPAL system) | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Change from baseline to 1 week and two weeks follow in motor symptoms as assessed with sensor recordings (OPAL system), movements will be recorded with digital sensors (gait and other tasks)

SECONDARY OUTCOMES:
Changing from baseline of measures from clinical scale (SARA) | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Changing from baseline of measures from clinical scale:
  SARA: Scale for the assessment and rating of ataxia
Changing from baseline of measures from clinical scale (ICARS) | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Changing from baseline of measures from clinical scale:
  ICARS: International cooperative ataxia rating scale
Changing from baseline of measures from clinical scale (UMSARS) | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Changing from baseline of measures from clinical scale:
  UMSARS: Unified multiple system atrophy rating scale
Changing from baseline of measures from patient related outcome | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Changing from baseline of measures from patient related outcome Euro 5 dimension quality of life (EQ5D)
Changing from baseline of measures from patient related outcome | Baseline (t0), at 1 week (t1), at 2 weeks (t2)
  Changing from baseline of measures from patient related outcome Clinical global impression (CGI)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per le Malattie Neurodegenerative (CEMAND) Dipartimento di Medicina e chirurgia, Sezione Neuroscienze, Università di Salerno, Salerno, Sa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Erro R, Antelmi E, Bhatia KP, Latorre A, Tinazzi M, Berardelli A, Rothwell JC, Rocchi L. Reversal of Temporal Discrimination in Cervical Dystonia after Low-Frequency Sensory Stimulation. Mov Disord. 2021 Mar;36(3):761-766. doi: 10.1002/mds.28369. Epub 2020 Nov 7. PMID 33159823
- [Background] Erro R, Tinazzi M, Morgante F, Bhatia KP. Non-invasive brain stimulation for dystonia: therapeutic implications. Eur J Neurol. 2017 Oct;24(10):1228-e64. doi: 10.1111/ene.13363. Epub 2017 Aug 7. PMID 28782903
- [Background] Datta A, Bansal V, Diaz J, Patel J, Reato D, Bikson M. Gyri-precise head model of transcranial direct current stimulation: improved spatial focality using a ring electrode versus conventional rectangular pad. Brain Stimul. 2009 Oct;2(4):201-7, 207.e1. doi: 10.1016/j.brs.2009.03.005. PMID 20648973